CLINICAL TRIAL: NCT02344017
Title: Safety and Pharmacokinetics of ODM-204 in Patients With Metastatic Castration-Resistant Prostate Cancer (CRPC): Open, Non-Randomised, Uncontrolled, Multicentre, Dose Escalation, First-in-man Study With a Dose Expansion
Brief Title: Safety and Pharmacokinetics of ODM-204 in Patients With Metastatic Castration-Resistant Prostate Cancer
Acronym: DUALIDES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3116001
Record Dates: First submitted 2014-12-29; First posted 2015-01-22 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ODM-204; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ODM-204 Phase I dose escalation (Experimental): Dose escalation
  Interventions: Drug: ODM-204; Drug: Prednisone
- ODM-204 Phase II dose expansion (Experimental)
  Interventions: Drug: ODM-204; Drug: Prednisone

INTERVENTIONS:
Drug: ODM-204 — co-administered with prednisone, orally daily
Drug: Prednisone — ODM-204 is co-administered with oral prednisone

SUMMARY:
The purpose of this first-in-man study is to evaluate safety, tolerability and pharmacokinetics of ODM-204 in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
The safety profile of ODM-204 will be explored together with the pharmacokinetics, pharmacodynamics and tumour response to treatment with ODM-204 to recommend the dosing regimen for further clinical studies. The pharmacokinetic properties of ODM-204 will be evaluated after single and multiple dose administrations at different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Male aged ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of prostate.
* Ongoing GnRH agonist or antagonist therapy, or after bilateral orchiectomy.
* Progressive metastatic disease
* Adequate bone marrow, hepatic, and renal function
* Acceptable and regular bowel movements without any GI disorder or procedure which may interfere with absorption of study treatment
* Ability to swallow study treatments

Exclusion Criteria:

* History of pituitary or adrenal dysfunction.
* Known brain metastases.
* Active infection or other medical condition that would make prednisone (corticosteroid) contraindicated.
* Uncontrolled hypertension
* Clinically significant heart disease
* Prolonged QTc interval

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by incidence of adverse events | Until disease progression, an expected average of 6 months
Safety and tolerability assessed by vitals signs and 12-lead ECG | Until disease progression, an expected average of 6 months
Safety and tolerability assessed by laboratory assessments | Until disease progression, an expected average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetic profile assessed by plasma peak concentration (Cmax) | 0 - week 12
Pharmacokinetic profile assessed by area under the concentration-time curve (AUC) | 0 - week 12
Pharmacokinetic profile assessed by time to reach peak concentration (tmax) | 0 - week 12
Preliminary antitumour activity assessed by prostate specific antigen (PSA) response | Until disease progression, an expected average of 6 months
Preliminary antitumour activity assessed by response in soft and bone tissues | Until disease progression, an expected average of 6 months
Pharmacodynamic profile assessed by hormone and circulating tumour cell measurements | 0 - week 12

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- Helsinki University Central Hospital, Helsinki, Finland
- Institut Gustave Roussy, Villejuif, France
- P. Stradins Clinical University Hospital, Riga, Latvia
- Velindre Cancer Centre, Cardiff, United Kingdom